CLINICAL TRIAL: NCT03979807
Title: The Role of Inhaler Device in the Treatment Persistence With Dual Bronchodilators in Patients With COPD
Brief Title: A Study Based on Medical Records That Looks at the Duration of Use of Two Types of Inhalers With Different Medicines in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0090
Record Dates: First submitted 2019-06-06; First posted 2019-06-07 (Actual); Results first posted 2020-07-23 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Tiotropium Bromide; GSK573719; vilanterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with Chronic obstructive pulmonary disease
  Interventions: Drug: Olodaterol/Tiotropium Bromide; Drug: Umeclidinium/ Vilanterol

INTERVENTIONS:
Drug: Olodaterol/Tiotropium Bromide — (Stiolto®) delivered via Respimat inhaler
Drug: Umeclidinium/ Vilanterol — (Anoro®) delivered via Ellipta Inhaler

SUMMARY:
To compare the persistence in using two different medications from the same drug class (LAMA/LABA FDC) which are delivered through different devices, a dry-powder inhalers (DPI) and Soft Mist Inhalers (SMI).

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Aged <40 years
* Enrolment with medical and pharmacy coverage prior to the cohort entry < 180 days
* Never had COPD diagnosis on the cohort entry date or prior to cohort entry
* A record for dispensed Olodaterol/Tiotropium Bromide delivered with Respimat inhalator or Umeclidinium/Vilanterol delivered with the Ellipta Inhaler during the 180-day baseline prior to cohort entry
* Diagnosis of asthma any time prior to cohort entry
* Diagnosis of lung cancer any time prior to cohort entry
* Diagnosis of lung transplant any time prior to cohort entry

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients initiating Olodaterol/Tiotropium Bromide or Umeclidinium/Vilanterol up to 2.5 years
Sampling Method: Non-Probability Sample
Enrollment: 11296 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aetion Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study compared the treatment persistence of patients with Chronic Obstructive Pulmonary Disease (COPD) using Olodaterol/Tiotropium Bromide inhaled via Respimat soft mist inhaler (SMI) versus patients with COPD using Umeclidinium/Vilanterol inhaled via the Ellipta Dry powder inhaler (DPI).
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included in the study. Initiators of Olodaterol/Tiotropium Bromide were matched to patients receiving Umeclidinium/Vilanterol using a 1:2 propensity score matching, resulting in a matched cohort of 11296 overall.
Groups:
- Olodaterol/Tiotropium Bromide - Matched Cohort: Propensity score matched cohort of patients with Chronic Obstructive Pulmonary Disease (COPD), who initiated Olodaterol/Tiotropium Bromide (Stiolto®) delivered with the Respimat soft mist inhaler (SMI), within the Truven MarketScan database between November 2015 and March 2018.
- Umeclidinium/Vilanterol - Matched Cohort: Propensity score matched cohort of patients with Chronic Obstructive Pulmonary Disease (COPD), who initiated Umeclidinium/Vilanterol (Anoro®) delivered with the Ellipta dry powder Inhaler (DPI), within Truven MarketScan database between November 2015 and March 2018.
Period: Overall Study
Arm/Group | Olodaterol/Tiotropium Bromide - Matched Cohort | Umeclidinium/Vilanterol - Matched Cohort
Started | 3876 | 7420
Completed | 3876 | 7420
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1:2 propensity score matched cohort of initators of Olodaterol/Tiotropium Bromide and Initiators of Umeclidinium/Vilanterol, identified from Truven MarketScan Claims database between November 2015 and March 2018.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olodaterol/Tiotropium Bromide - Matched Cohort | Umeclidinium/Vilanterol - Matched Cohort | Total
Number analyzed (Participants) | 3876 | 7420 | 11296
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.63 (10.50) | 64.58 (10.53) | 64.60 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1785 | 3409 | 5194
  Male | 2091 | 4011 | 6102
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Rate of Discontinuation of Index Treatment (Olodaterol/Tiotropium Bromide or Umeclidinium/Vilanterol)
Description: The primary outcome of interest was discontinuation of index treatment (Olodaterol/Tiotropium Bromide or Umeclidinium/Vilanterol), defined as persistence, (i.e. no refill Claim within 60 days [not including treatment Switch, nor death] after end of supply) during follow-up. Persistence was assessed by calculating rates of discontinuation in the matched cohorts using a 60-day allowable gap. Rates of discontinuation are reported as the number of events divided by the number of Person-years at risk. Addition of another treatment to index treatment did not count as discontinuation.
Time Frame: From first day after the cohort entry date to the earliest occurence of the outcome (discontinuation or refills), or any censoring criteria (365 days of follow-up without discontinuation, death, disenrollment end of data).
Population: 1:2 propensity score matched cohort of initiators of Olodaterol/Tiotropium Bromide and initiators of Umeclidinium/Vilanterol, identified from Truven MarketScan Claims database between November 2015 and March 2018.
Measure: Number; unit: Events per 1000 person-years
Arm/Group | Olodaterol/Tiotropium Bromide - Matched Cohort | Umeclidinium/Vilanterol - Matched Cohort
Number analyzed (Participants) | 3876 | 7420
Events per 1000 person-years | 1826.00 | 1647.03
Statistical Analysis 1: Comparison: Olodaterol/Tiotropium Bromide - Matched Cohort vs Umeclidinium/Vilanterol - Matched Cohort; Test type: Other; Adjusted Hazard Ratio = 1.11, 95% CI 2-sided [1.06 to 1.17] — Cox proportional hazard model. 'Treatment' is the only Independent variable used to estimate the hazard ratios. Umeclidinium/Vilanterol is Reference Group

ADVERSE EVENTS:
Description: As this is a non-interventional study with secondary use of data retrieved from a US health claims database, safety monitoring and safety reporting on an individual case level is not applicable.
Arm/Group | Olodaterol/Tiotropium Bromide - Matched Cohort | Umeclidinium/Vilanterol - Matched Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
By using data from insurance claims, data are based on a large, non-random convenience sample, which may contain biases or lack generalizability to other populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT03979807/Prot_SAP_000.pdf